CLINICAL TRIAL: NCT01620723
Title: Effect Evaluation of a Theory and Evidence Based Programme for Establishing Effective Breastfeeding After Short Time Hospitalization Post Partum
Brief Title: Evaluation of Breastfeeding Support After Short Time Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Committee for Health Education (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Ingrid Nilsson, Senior Project Coordinator, Danish Committee for Health Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7111442
Record Dates: First submitted 2012-06-12; First posted 2012-06-15 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; Breastfeeding self efficacy
MeSH Terms: conditions — Breast Feeding | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New breastfeeding programme (Experimental): The breastfeeding programme consists of four core elements:
  1. breastfeeding is a parental task
  2. skin to skin contact during the first three days
  3. frequent breastfeeding at least 8 times a day
  4. good positioning, preferable in a laid back position
  Moreover communication was supposed to enhance breastfeeding self-efficacy, using Banduras theory of self-efficacy
  Interventions: Other: New Breastfeeding Counselling
- Treatment as usual (Active Comparator): Breastfeeding counselling uses the national handbook of breastfeeding as reference
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: New Breastfeeding Counselling — An intervention will be developed during the first part of the study. The intervention is supposed to consist of evidence based actions to support the metabolic adaptation of the newborn, establishment of the milk production of the mother and increase the breastfeeding self efficacy of the mother.
  Arms: New breastfeeding programme
Other: Treatment as usual — Health professionals offer the usual care for the breastfeeding mother
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is to evaluate if the developed theory and evidence based programme has a positive effect on mother's breastfeeding self efficacy, establishing an effective breastfeeding and breastfeeding duration after short time hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women (gestational week 35-36)

Exclusion Criteria:

* women with known physical, psychological and/or social illness/problem that result in hospitalization more than 50 hours after delivery
* women with known pregnancy related illness that result in hospitalization more than 50 hours after delivery
* Women not understanding or speaking Danish
* women expecting multiple babies
* women having decided not to breastfeed
* women expecting to deliver at another hospital than the one she has been visiting during pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3541 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Parents breastfeeding self efficacy | 7 days post partum

SECONDARY OUTCOMES:
Effective breastfeeding | 7 days post partum
  Effective breastfeeding is measured by the outcome measures: breastfeeding frequency, milk coming in before 3rd day pp, number of stools 3 days pp, baby's swallowing of milk
Duration of exclusive and full breastfeeding | 7 and 30 days post partum and 6 month post partum
Baby's morbidity | 7 and 30 days post partum and 6 month post partum
  Measuring jaundice, dehydration, use of health facilities
Breastfeeding problems | 7 and 30days and 6 month post partum
  Measuring nipple pain and fissures, too much or too little milk

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Nilsson, RN, MSA, IBCLC, Principal Investigator — Danish Committee for Health Education
Locations (9):
- Denmark (9):
  - Aalborg Sygehus, Aalborg
  - Sygehus Vendsyssel, Hjørring
  - Horsens sygehus, Horsens
  - Kolding Sygehus, Kolding
  - Nykøbing F Sygehuse, Nykøbing Falster
  - Regionshospitalet Randers, Randers
  - Haderslev/Sønderborg sygehus, Sønderborg
  - Sygehus Thy-Mors, Thisted
  - Regionshospitalet Viborg, Viborg

REFERENCES:
- [Derived] Yonemoto N, Nagai S, Mori R. Schedules for home visits in the early postpartum period. Cochrane Database Syst Rev. 2021 Jul 21;7(7):CD009326. doi: 10.1002/14651858.CD009326.pub4. PMID 34286512